CLINICAL TRIAL: NCT05203107
Title: Cross-cultural Adaptation of Urdu Version of Menstrual Attitude Questionnaire: A Reliability and Validity Study
Brief Title: Urdu Version of Menstrual Attitude Questionnaire: A Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-0272
Record Dates: First submitted 2021-10-26; First posted 2022-01-24 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Menstruation
Keywords: Attitude; Menstruation; females; psychometric properties; Menstrual Attitude Questionnaire
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the validity and reliability of Urdu version of Menstrual Attitude Questionnaire

DETAILED DESCRIPTION:
Menstrual Attitude Questionnaire has been distributed in 200 women who were recruited by convenience sampling technique under the pre defined inclusion and exclusion criteria after signing the informed consent forms .

This study's findings will assist determine the Menstrual Attitude Questionnaire's reliability and validity in individuals with neck pain and impairment. This scale's reliability will be evaluated utilising internal consistency and test-retest methods. Cronbach's alpha value checks internal consistency. The interclass correlation will be used to examine the test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

1. A history of lower abdominal pain for more than 6 menstrual cycle.
2. No elective treatment counting TENS inside 1 month earlier to enrollment within the ponder.
3. Provision of informed consent prior to enrollment in the study.

Exclusion Criteria:

1. Pregnant or Breastfeeding
2. History of surgery of the lower abdomen.
3. Heart disease.
4. Cancer.
5. Severe mental disorder

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females of 18-36 years of age group
Study Population: Pregnant or Breastfeeding Women
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Menstrual attitude questionnaire(MAQ) | 1st day
  Menstrual Attitude Questionnaire Performa positive and negative items are scored in a 7 point Likert scale. Larger the score, higher is the level of agreement with the issued targeted. Range of score starts from 1 (strongly disagree) to 7 (strongly agree). Since then, Menstrual Attitude Questionnaire has been used in many studies among various populations in various races and nations. It can be used in the assessment of individuals situations related to menstruation. The investigators have translated this questionnaire into Urdu and 200 females were participated in this study.
Beliefs about and Attitudes toward Menstruation Questionnaire | 1st day
  Beliefs about and Attitudes toward Menstruation Questionnaire is a 5-point Likert scale questionnaire designed to access the belief and attitudes towards the menstrual cycle of the female gender. It has 45 questions with 5 options from strongly disagree to strongly agree. Various attitudes related to various stages of the menstrual cycle and related myths and false beliefs are accessed. The investigators used this questionnaire to evaluate the attitudes and beliefs of the females of attending various hospital of our city.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No